CLINICAL TRIAL: NCT00730834
Title: Phase 4 Study of Use of a Customized Acoustic Stimulus to Reduce the Disturbing Symptoms of Tinnitus and Hyperacusis
Brief Title: Customized Acoustic Stimulation for Long Term Medical Benefit for the Relief of Tinnitus and Hyperacusis
Acronym: CALM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neuromonics, Inc. (Industry)
Responsible Party: Jack Wazen, MD, Silverstein ear institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALM Study; 20071022
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Tinnitus; Hyperacusis
Keywords: tinnitus; ringing in the ears; buzzing; static; hyperacusis; loudness discomfort; Clinically; significant; discomfort
MeSH Terms: conditions — Tinnitus; Hyperacusis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Oasis — Digital sound player that provides customized acoustic stimulus based on subjects hearing thresholds
  Other Names: Neuromonics Oasis Tinnitus Treatment

SUMMARY:
Neuromonics TInnitus Treatment CALM study is a multi site study of 100 adult subjects with clinically significant disturbing tinnitus to evaluate outcome measures using the FDA cleared Neuromonics treatment after 6, 12, 24 and 36 months. Patients must be meet certain inclusion criteria and they are also required to pay for the all costs of the treatment. Subjects will be provided a modest participation fee at 6, 12, 24 and 36 months upon completion of patient questionnaires (subjects must have access to a computer and internet in order to complete on line questionnaires).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age,
* TRQ of at least 17 or above,
* Able to pay for the treatment,
* Not using any other treatment for tinnitus,
* Access to computer and internet,
* Compliant patient

Exclusion Criteria:

* Hearing PTA > 50 dB, score on HADS of greater than 11 on the anxiety and depression scale,
* Not willing to follow the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-06; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Pre and post treatment scores on Tinnitus reaction questionnaire | 6, 12, 24, 36 months

SECONDARY OUTCOMES:
Tinnitus Handicap Inventory, Hospital Anxiety and Depression Scale, | 6, 12, 24, 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Silverstein Ear Institute, Sarasota, Florida, United States

REFERENCES:
- See also: Related Info — http://www.neuromonics.com